CLINICAL TRIAL: NCT06769139
Title: Evaluation of the Impact of Red Blood Cell Exchange on Thrombo-inflammation in Sickle Cell Disease STIREX : Sickle Cell Disease - Thrombo-Inflammation - Red Blood Cell EXchange
Brief Title: Evaluation of the Impact of Red Blood Cell Exchange on Thrombo-inflammation in Sickle Cell Disease
Acronym: STIREX
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0509
Record Dates: First submitted 2024-11-18; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease
Keywords: thrombo-inflammation; Red blood cell Exchange
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sickle patients treated by red blood cell exchange: 20 adult sickle cell patients treated by red blood cell exchange (10 patients on manual exchange and 10 patients on automatized exchange)
  Interventions: Other: Red blood cell exchange

INTERVENTIONS:
Other: Red blood cell exchange — Red blood cell exchange manual exchange and automatized exchange

SUMMARY:
Sickle cell disease is the most common inherited blood disorder worldwide. It is a hemoglobinopathy characterized by chronic hemolysis, endotheliopathy, coagulation activation, and chronic inflammation. It is a multisystemic disease leading to acute (vaso-occlusive crisis, acute chest syndrome, stroke…) and chronic complications with multiorgan damage. Thrombo-inflammation is defined by the cooperation and interaction between hemostasis and the innate immune system. The platelet represents the cornerstone of this phenomenon, being at the interface of these two systems. In sickle cell disease, platelets are activated and release cytokines, leading to a pro-coagulant and pro-inflammatory state. Transfusion, whether occasional or chronic, is a major sickle cell disease treatment. It is common to distinguish simple transfusion from exchange transfusion. The latter involves replacing a given volume of sickle red blood cells with healthy red blood cells. Exchange transfusion allows avoiding an excessive increase in hemoglobin. The decrease of hemoglobin S under 30% achieved by red blood cell exchange reduces the risk of stroke by more than 90% in children with cerebral vasculopathy. Moreover, transfusion can be used in acute complications such as vaso-occlusive crisis and acute chest syndrome. Despite this efficacy, a subgroup of patients is not totally protected against acute and chronic complications. The persistence of chronic inflammation is suggested. To date, it is not known if red blood cell exchange can reduce the thrombo-inflammatory dynamic in sickle cell disease. The aim of this study is to evaluate the impact of red blood cell exchange on thrombo-inflammatory parameters in 20 adult sickle cell patients (10 patients on manual exchange and 10 patients on automatized exchange).

DETAILED DESCRIPTION:
Prospective observational cohort with additional blood samples. This study is monocentric.

ELIGIBILITY:
Inclusion Criteria:

* Sickled Cell Disease patient with SS or S/beta thalassemia genotype
* Red blood cell exchange > 3 months
* Up-to-date social security coverage
* Patient able to understand the purpose and constraints of the research project
* Patient has read the study information leaflet and does not object to the research.

Exclusion Criteria:

* Thrombopenia < 50 G/L
* Non-steroidal anti-inflammatory drugs < 7 days before enrolment
* Anti-platelet agents < 7 days before enrolment
* Pregnancy or breastfeeding
* Patient objects to take part in the study
* Patient under guardianship, curatorship or safeguard of justice
* Patients with ongoing clinical trial requiring collection of additional blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified during a follow-up consultation in the internal medicine department.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of thrombo-inflammation parameters in sickle patients treated by red blood cell exchange | 2 days
  Thrombo-inflammation is evaluate using a composite criteria composed by 4 thromo-inflammatory parameters : soluble platelet activation markers, inflammasome, platelet response, circulating platelet microparticles and lipidomic study of plasma eicosanoids.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre COUGOUL, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Oncopole - Toulouse Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided